CLINICAL TRIAL: NCT02690831
Title: Effects of Manual Therapy and Respiratory Muscle Training on the Maximal Inspiratory Pressure in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Pablo Candelas Fernández, Physiotherapist, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad Autonoma de Madrid
Record Dates: First submitted 2015-12-16; First posted 2016-02-24 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Manual Therapies; Respiratory Muscle Training; Exercise Therapy; Inspiratory Capacity; Asthma
Keywords: Asthma; Inspiratory Muscle Training; Manual Therapies
MeSH Terms: conditions — Asthma | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Inspiratory Muscle training (IMT) (Active Comparator): The IMT program consisted of supervised and domiciliary exercises:
  1. - The supervised exercises was performed in the presence of physiotherapist. This consisted of 30 min 2 days for 6 weeks using the threshold device (Powerbreathe classic level 1, Gaiam Ltd; Southam, Warwickshire, UK). This program involve 5 sets of 5 repetitions with 30 seconds rest between each one. The load of the training was distributed as follow:
     * First week: 30% Maximum Inspiratory Pressure (MIP)
     * Second week: 40% MIP
     * Third week: 50% MIP
     * Fourth week: 50% MIP
     * Fifth week: 60% MIP
     * Sixth week: 60% MIP
  2. - The domiciliary exercises consisted of Yoga Breathing Exercises (Pranayama) that combines the inspiration and expiration through one or both nostrils, and requires the activation of chest and abdomen.
  Interventions: Other: Inspiratory Muscle training (IMT); Device: Powerbreathe
- IMT + Manual Therapy and Motor Control Exercise (Experimental): The protocol for this group is identical to the previous group with the sole difference that is added a manual therapy (MT) and a motor control exercises (MCE). The MT protocol was performed for 15min, whereas the MCE was 10min. Below it described both protocols:
  1. - MT:
     * Upper cervical region mobilization in flexion
     * Lower cervical postero-anterior mobilization + maintained traction
     * Costovertebral joint postero-anterior mobilization
     * Thrust dorsal
     * Cervical postero-anterior mobilization
  2. - MCE:
     * Isometric contraction of the deep neck flexors.
     * Isometric contraction of the neck extensors.
     * Neural self-mobilization.
     * Cervical retraction with theraband.
     * Sphinx.
     * Scapular adduction exercises in prone.
     * Scapular adduction exercises in sitting position with theraband.
  Interventions: Other: IMT + Manual Therapy and Motor Control Exercise; Device: Powerbreathe

INTERVENTIONS:
Other: Inspiratory Muscle training (IMT) — Inspiratory Muscle training This protocol will be performed using the Powerbreathe classic level 1 device and Yoga Respiratory Exercises (Pranayama)
  Arms: Inspiratory Muscle training (IMT)
Other: IMT + Manual Therapy and Motor Control Exercise — IMT + Manual Therapy and Motor Control Exercise The Inspiratory Muscle Training protocol will be performed using the Powerbreathe classic level 1 device and Yoga Respiratory Exercises (Pranayama). Manual Therapy and Motor Control Exercises will consist of joint mobilization/manipulation and exercises in the neck and thoracic regions
  Arms: IMT + Manual Therapy and Motor Control Exercise
Device: Powerbreathe

SUMMARY:
The aim of this study is to assess if an intervention of manual therapy and motor control exercises combined with an inspiratory muscle training program is more effective than an inspiratory muscle training program alone in increasing the maximum inspiratory pressure in patients with asthma. In addition, the study pretends to evaluate the changes caused by the intervention regarding possible postural changes and thoracic diameter.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatics subjects aged between 18 and 65 years

Exclusion Criteria:

* Were excluded participants who presented neurologic, psychiatric or cognitive pathologies which difficult the cooperation, inflammatory disease of the cervical spine and/or severe orthopedic problems that difficult the daily activities, history of thoracic surgery, vertebral fracture, abnormal thorax radiography, spinal and thoracic structured musculoskeletal disorders and to present any contraindication of treatment techniques (e.g. ostheophorosis). In case of exacerbation of asthma, missing more than one treatment session and/or to appear any contraindication to continue the treatment routine during the six weeks of the study the patient also were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure | Change from Baseline in Maximum Inspiratory Pressure at 6 weeks
  The maximum inspiratory pressure (MIP) was measured with a device called Kinetic KH1 Powerbreath in cmH2O. This device applies an inspiratory load which provides a resistance. The maneuver was performed in a sitting position. Measuring a minimum of 3 times was performed, recording the highest value

SECONDARY OUTCOMES:
Head posture | Change from Baseline in Head Posture at 6 weeks
  The head posture was measured through the Cervical Range of Motion (CROM) device in centimetres. This instrument measures physiological movements of the cervical spine and head position. It´s a reliable method of measuring, providing a range of intra-meter reliability from 0.7 to 0.9 and a range of inter-meter reliability from 0.8 to 0.87. The evaluator instructed the patient to sit in a standardized position and assume a natural position of the head and the goniometer was placed over his head to measure the head posture.
Thoracic kyphosis | Change from Baseline in Thoracic kyphosis at 6 weeks
  The measurement of the thoracic kyphosis was performed through flexicurve in degrees. It is a flexible rule that is molded to the back of the subject in order to replicate the shape of the spine. The flexicurve is a valid and reliable tool. The spinous processes of C7 and T12 were located, subsequently it placed on paper 10x10 to draw the curve and to obtained the index flexicurve.
Forced Vital Capacity (FVC) | Change from Baseline in Volumes and lung capacities at 6 weeks
  The measurement of the Forced Vital Capacity was performed through a simple Spirometry.The Spirometry was performed according to American Thoracic Society criteria and was measured in litres. The maneuver was performed 3 times and recording the best one.
Forced Expiratory Volume at the First second (FEV1) | Change from Baseline in Volumes and lung capacities at 6 weeks
  The measurement of the Forced Espiratory Volumen at first second was performed through a simple Spirometry.The Spirometry was performed according to American Thoracic Society criteria and was measured in litres. The maneuver was performed 3 times and recording the best one.
Peak Expiratory Flow (PEF) | Change from Baseline in Volumes and lung capacities at 6 weeks
  The measurement of the Peak Expiratory Flow was performed through a simple Spirometry.The Spirometry was performed according to American Thoracic Society criteria and was measured in litres. The maneuver was performed 3 times and recording the best one.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Superior de Estudios Universitarios La Salle, Madrid, Madrid, Spain